CLINICAL TRIAL: NCT00479518
Title: Prognostic Value of Cardiac and Renal Markers in the Acute Phase of Ischemic Stroke or Transient Ischemic Attack :Albuminuria-Brain Natriuretic Peptide-Cystatine C in Stroke
Brief Title: Prognostic Value of Cardiac and Renal Markers in Ischemic Stroke and Transient Ischemic Attack
Acronym: ABC-AVC
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHRI06-IB Cohorte ABC-AVC
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: stroke; transient ischemic attack; albuminuria; BNP; Cystatin C
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Stroke; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with stroke or transient ischemic attack (TIA) are at high risk of poor outcome, recurrence of cardiovascular events or vascular death.Until now, no reliable predictive biological marker could be identified in the acute phase of stroke.We hypothese that, in the acute phase of ischemic stroke or TIA, the increase of cardiac ( brain natriuretic peptide, BNP) or renal markers (albuminuria, cystatin C)might predict recurrence of cardiovascular events or vascular death. We want to assess which one of these markers has the best prognosis value , in a prospective study of 300 stroke patients followed during 3 years.

DETAILED DESCRIPTION:
Patients with ischemic stroke or TIA will be included in the 48 hours following the onset of symptoms, in 3 university hospitals.For each patient will be collected

* 1 blood sample for the BNP measure in pg/ml
* 1 blood sample for the Cystatin C measure in mg/l
* 2 urinary samples to measure the albumine/creatinine ratio, at inclusion and 5 days after the inclusion, and to study the variation of albuminuria in micrograms/min.

The clinical follow-up will be organized during 3 years. The following events will be notified: poor outcome (defined with the Barthel and Rankin scores), recurrence of cardiovascular or cerebrovascular events, vascular death.

After adjustment on the main clinical prognosis factors, we want to determine wich one of these markers has the best prognosis significance and allows to identify in the acute phase the "high-risk" patients, in order to intensify individual treatment and secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or TIA in the first 48 hours following the onset of symptoms

Exclusion Criteria:

* Patient unable to give an informed consent
* Urinary sample impossible to collect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Ischemic stroke or TIA
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BONNAUD Isabelle, MD, Principal Investigator — Service de Neurologie / CHRU de Tours
Locations (3):
- France (3):
  - Service de Neurologie / Hopital LAENNEC, Nantes
  - Service de neurologie / CHU Pontchaillou, Rennes
  - Service de Neurologie / CHRU de Tours, Tours